CLINICAL TRIAL: NCT06738901
Title: A Phase 1/3, Open-label, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of Human Plasma-derived Factor VIII (SKP-0141) for the Treatment and Prophylaxis in Male Patients with Severe Hemophilia a
Brief Title: An Open-label Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of SKP-0141 for the Treatment and Prophylaxis in Severe Hemophilia a Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SK Plasma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SKP-0141_HemA_I/III_2024
Record Dates: First submitted 2024-12-08; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hemophilia A, Severe
Keywords: Congenital hemophilia A; Prophylaxis; On-demand; FVIII concentrate; Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prophylactic treatment (Experimental)
  Interventions: Biological: SKP-0141

INTERVENTIONS:
Biological: SKP-0141 — Human plasma-derived coagulation factor VIII concentrate

SUMMARY:
This is a prospective, multicenter, open-label study to assess efficacy, safety, pharmacokinetics (PK), and immunogenicity of human plasma-derived Factor VIII (FVIII) in previously treated patients (PTPs) with severe hemophilia A. Overall, 55 male PTPs aged 12 to 65 years old with a FVIII level of < 1% and at least 150 treatment exposure days (EDs) with a previous FVIII product will be enrolled. Patients will receive SKP-0141 at a dose of 25 to 50 IU/kg every second day or 3 times per week for at least 50 EDs and/or 6 months from the start of prophylactic treatment. Efficacy of SKP-0141 will be primarily evaluated in bleeding prophylaxis with annualized bleeding rate from start of treatment and until end of treatment (Visit 10).

ELIGIBILITY:
Inclusion Criteria:

* A patient or parent/legal guardian who is capable of giving signed informed consent
* Patients assigned male at birth and must be 12 to 65 years old at the time of Screening
* Diagnosis of severe congenital hemophilia A, defined as an FVIII level of <1% as documented in the patient's medical records at the time of Screening
* Patients who have received or are currently receiving plasma-derived and/or recombinant FVIII products and have had at least 150 EDs with a FVIII product
* Patients who can produce viable sperm and have a partner of childbearing potential must agree to take appropriate contraceptive measures consistently during the study, starting at Screening and until 30 days after the end of study

Exclusion Criteria:

* Any history of or current FVIII inhibitors or any first order family history of FVIII inhibitors in terms of detectable FVIII inhibitors (ie, ≥0.6 Bethesda Units [BU]) using the Nijmegen-modification of the Bethesda assay
* Any known congenital or acquired coagulation disorder other than the congenital hemophilia A
* Evidence of thrombosis, including deep vein thrombosis, stroke, pulmonary embolism, myocardial infarction, and arterial embolus within 3 months prior to Visit 1
* Experienced life-threatening bleeding episode or had major surgery or an orthopedic surgical procedure during the 3 months prior to Visit 1
* Has been tested positive for HIV with a CD4+ count ≤200/μL at Screening (if available, hepatitis B surface antigen, or hepatitis C virus antibodies, and/or positive hepatitis B virus deoxyribonucleic acid/HCV ribonucleic acid at Screening
* Platelet count <100 000/μL at Screening
* Patients with serum aspartate aminotransferase or serum alanine aminotransferase values >5 × the upper limit of normal or serum creatinine values >2 × ULN at Screening
* Patients who are currently receiving IV immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment within 3 months prior to Visit 1
* Use of any other investigational medicinal product, cryoprecipitate, whole blood, or plasma within 30 days or 5 half-lives prior to Visit 1
* Known or suspected hypersensitivity to any FVIII product or their excipients
* Has a physical, medical, or psychological condition, that in the opinion of the PI, may interfere with the evaluation of the study.
* Are study site personnel directly affiliated with this study and their immediate families

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate | Up to 25 weeks
  Efficacy of SKP-0141 in bleeding prophylaxis in previously treated patients with severe hemophilia A based on the number of bleeding episodes per year

SECONDARY OUTCOMES:
Hemostatic response | Up to 25 weeks
  Efficacy of SKP-0141 for the treatment of breakthrough bleeding episodes using a 4-point scale in previously treated patients with severe hemophilia A
Consumption of SKP-0141 required for prophylaxis | Up to 25 weeks
  Dose of SKP-0141 injections (IU/kg/year and IU/kg/month) required for prophylaxis in previously treated patients with severe hemophilia A
Consumption of SKP-0141 required for on-demand treatment | Up to 25 weeks
  Dose/number of SKP-0141 injections (IU/kg/bleed) required for treatment of bleeding episodes in previously treated patients with severe hemophilia A
Peak plasma concentration (Cmax) | At 1 week and 25 weeks
  Maximum plasma concentration of SKP-0141 in previously treated patients with severe hemophilia A
Time to reach peak plasma concentration (Tmax) | At 1 week and 25 weeks
  Time to reach peak plasma concentration of SKP-0141 in previously treated patients with severe hemophilia A
Area under the plasma concentration versus time curve (AUC) | At 1 week and 25 weeks
  Area under the plasma concentration versus time curve in previously treated patients with severe hemophilia A
Half-life (T1/2) | At 1 week and 25 weeks
  Half-life of SKP-0141 in previously treated patients with severe hemophilia A
Total plasma clearance (CL) | At 1 week and 25 weeks
  Total plasma clearance of SKP-0141 in previously treated patients with severe hemophilia A
Elimination constant (Kel) | At 1 week and 25 weeks
  Elimination rate constant of SKP-0141 in previously treated patients with severe hemophilia A
Volume of distribution (Vd) | At 1 week and 25 weeks
  Volume of distribution of SKP-0141 in previously treated patients with severe hemophilia A
Mean residence time (MRT) | At 1 week and 25 weeks
  Mean residence time in vivo of SKP-0141 in previously treated patients with severe hemophilia A
Incremental in vivo recovery (IVR) | At 1 week and 25 weeks
  Incremental in vivo recovery (IVR) in previously treated patients with severe hemophilia A
Incidence of treatment-emergent adverse events (TEAEs) | Up to 26 weeks
  Incidence of treatment-emergent adverse events in previously treated patients with severe hemophilia A
Incidence of serious adverse events (SAEs) | Up to 26 weeks
  Incidence of serious adverse events in previously treated patients with severe hemophilia A
Incidence of adverse events of special interest (AESIs) | Up to 26 weeks
  Incidence of adverse events of special interest in previously treated patients with severe hemophilia A
Incidence of adverse events (AEs) | Up to 26 weeks
  Incidence of adverse events in previously treated patients with severe hemophilia A
Incidence of clinically significant changes | Up to 25 weeks
  Safety and tolerability of SKP-0141 in previously treated patients with severe hemophilia A based on the incidence of clinically significant changes from baseline in safety laboratory evaluations (hematology, serum chemistry, and urinalysis), vital signs (pre- and post-injection), physical examinations, and ECG
Incidence of FVIII inhibitor formation | Up to 25 weeks
  Immunogenicity of SKP-0141 from incidence of FVIII inhibitor formation (≥0.6 Bethesda Units) calculated using the Nijmegen-modified Bethesda assay in previously treated patients with severe hemophilia A

OTHER OUTCOMES:
Hemostatic response in surgical prophylaxis | Perioperatively/Periprocedurally
  Hemostatic response (efficacy) of SKP-0141 in surgical prophylaxis in previously treated patients with severe hemophilia A

IPD SHARING:
Plan to Share IPD: No